CLINICAL TRIAL: NCT04130711
Title: Preliminary Study to Evaluate the Effect of an EEG-proprioceptive Neurofeedback on Cortical Excitability and Motor Function of the Upper Limb After Stroke
Brief Title: HAptic Neurofeedback Design for Stroke
Acronym: HANDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC19_8866_HANDS
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: stroke; neurofeedback; tendon vibration; virtual reality; haptic
MeSH Terms: conditions — Stroke | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TEST 1: Visual virtual Conditions (Other): * 50 subjects (30 healthy volunteers and 20 patients after stroke)
  * 3 different situations of vibration applications, without EGG neurofeedback session
  Interventions: Other: Visual virtual Conditions
- TEST 2: Standard EEG (Other): * 20 subjects (healthy volunteers)
  * 3 separate electroencephalographic recording conditions without Neurofeedback
  Interventions: Other: Standard EEG
- TEST 3: Neurofeedback Training Stroke Patients (Other): * 26 patients after stroke
  * 12 neurofeedback sessions spread over 6 weeks according to the feedback modality that will be drawn (visual or visuo-vibratory)
  Interventions: Other: Neurofeedback Training Stroke Patients

INTERVENTIONS:
Other: Visual virtual Conditions — The objective is to evaluate if certain virtual visual conditions can increase the illusion of movement induced by the tendon vibration of the upper limb.
  Thirty healthy volunteers and 20 post-stroke subjects will test 3 different situations of vibration applications, with no EEG Neurofeedback session. It will be applied to the subject (healthy and post-stroke) according to a randomized order a vibrator for a few minutes on his non-dominant (or deficit) hand hidden from view, with a screen representing a static virtual hand, then a vibrator on his hand hidden with a screen representing an animated virtual hand, then a vibrator on his hand hidden with a screen representing an empty background.
  Other Names: 3 different situations of vibration applications, without EGG neurofeedback session
  Arms: TEST 1: Visual virtual Conditions
Other: Standard EEG — Twenty healthy volunteers test 3 separate electroencephalographic recording conditions without Neurofeedback. It will be applied to the subject an EEG headset recording brain activity during the application of vibration stimulation producing the illusion of movement on the non-dominant hand or during a task Mental imagery of the upper limb, or during the joint application of vibratory stimulation and a mental imaging task on the affected upper limb in a randomized order.
  Other Names: 3 separate electroencephalographic recording conditions without Neurofeedback
  Arms: TEST 2: Standard EEG
Other: Neurofeedback Training Stroke Patients — The post-stroke subject is evaluated on clinical tests (FMA, ARAT, MAL, NHPT, Finger Tapping test) during the first visit. Then, he performs 12 sessions of NFB (on his deficit member) lasting 45 minutes, spread over 6 weeks, depending on the feedback modality that has been drawn randomly (visual or visuo-vibratory). A second visit after the first NFB session and a third visit after the last NFB session evaluates the motor skills of the trained upper limb (FMA, ARAT, MAL, NHPT, Finger Tapping test) and a satisfaction questionnaire is given to the subject for evaluate tolerance and satisfaction with the feedback modality assigned. Evaluation of changes of EEG sensorimotor rhythms at the end of the program.
  Other Names: 12 neurofeedback sessions spread over 6 weeks according to the feedback modality that will be drawn (visual or visuo-vibratory)
  Arms: TEST 3: Neurofeedback Training Stroke Patients

SUMMARY:
Interventional study with minimal risks and constraints, prospective, monocentric.

DETAILED DESCRIPTION:
Many patients with stroke have a severe motor deficit in the upper limb impacting their independence. Electroencephalogram (EEG) Neurofeedback is a re-education technique that improves cerebral plasticity and motor gain in these people during the chronic phase of stroke. The visual feedback usually used tends to diminish the subject's attentional resources, while the proprioceptive feedbacks appear to be more effective on cortical excitability. Vibration feedback inducing movement illusion has been shown to be effective in healthy subjects, but has not been tested in people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers : Major (age greater than or equal to 18 years) and under 80 years; Free, informed and written consent signed by the volunteer; Absence of clinical neurological antecedents that can interact with the achievement of the motor task or with the EEG signal.
* Patients after stroke : Major (age greater than or equal to 18 years) and under 80 years;Ischemic or unilateral cerebral hemorrhagic hemorrhagic attack;Stroke dating back more than 6 months (considered as a delay where recovery of the upper limb to wait is less with conventional rehabilitation);Mild to severe upper limb deficiency: FMA-EU score ≤ 60; Free, informed and written consent signed by the patient or a member of his entourage (in the case of a patient able to understand the information and to express his / her consent but presenting motor difficulties leading to an invalid signature).

Exclusion Criteria:

* Healthy Volunteers : major persons subject to legal protection, persons deprived of their liberty
* Patients after stroke : Ischemic or hemorrhagic involvement of posterior fossa (brainstem, cerebellum);Complete motor deficiency of the upper limb (FMA-UE = 0);Epicritic and proprioceptive anesthesia;Understanding difficulties limiting participation in the study;Major persons subject to legal protection, persons deprived of their liberty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Relative Power of Event Related Desynchronization in µ et beta EEG bands of healthy controls and stroke participants | throught study completion, in the 5th week after the onset of the experiment for each participant
  The relative increase of Event Related Desynchronization (ERD) relative power sensorimotor rhythms (µ et beta bands) in EEG during the last session of NeuroFeedBack in the motor cortex, between motor imagery and rest, measured in microvolt

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie COGNE, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Derived] Le Franc S, Bonan I, Fleury M, Butet S, Barillot C, Lecuyer A, Cogne M. Visual feedback improves movement illusions induced by tendon vibration after chronic stroke. J Neuroeng Rehabil. 2021 Oct 30;18(1):156. doi: 10.1186/s12984-021-00948-7. PMID 34717672